CLINICAL TRIAL: NCT01044472
Title: Multi-site Left Ventricular (MSLV) Pacing With Quartet 1458Q Lead
Acronym: MSLV
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-09-048-EU-HF
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Multi-site Left Ventricular Pacing
Keywords: CRT-D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and hemodynamic performance of the MSLV Pacing feature in a clinical setting.

DETAILED DESCRIPTION:
To evaluate the hemodynamic impact of different pacing MSLV configurations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a recognised indication to receive a CRT-D device or an upgrade from a pacemaker or ICD to a CRT-D system.
* Patients have signed an informed consent form indicating their willingness to participate to this study.

Exclusion Criteria:

* Patients who are unable to comply with the follow-up schedule based on their geographic location or for any reason.
* Patients with second or third degree AV Block
* Patients with intrinsic atrial rhythm < 40 bpm
* Patients with a previously implanted left ventricular pacing lead.
* Patients who are pregnant.
* Patients currently participating in a clinical investigation that includes an active treatment arm.
* Patients under 18 years of age.
* Patients with a life expectancy of less then 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard CRT-D indications
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (7):
  - Herzzentrum, Bad Krozingen
  - Kerckhoff - Klinik, Bad Nauheim
  - Herz-und Diabetes Zentrum NRW, Bad Oeynhausen
  - Schüchtermannklinik, Bad Rothenfelde
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt
  - Städt. Klinikum, Ludwigshafen
  - Klinikum Rosenheim, Rosenheim
- United Kingdom (3):
  - Russells Hall, Dudley
  - Liverpool Heart and Chest Hospital, Liverpool
  - St Thomas, London

IPD SHARING:
Plan to Share IPD: No